CLINICAL TRIAL: NCT07103642
Title: EXACERBATIONS AND REAL-WORLD OUTOMES INCLUDING CARDIOPULMONARY EVENTS AMONG PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE INITIATING BUDESONIDE/GLYCOPYRRONIUM/FORMOTEROL (MITOS: EROS+CP Japan Study)
Brief Title: EXACERBATIONS AND REAL-WORLD OUTOMES AMONG PATIENTS WITH COPD INITIATING BREZTRI (EROS+CP Japan Study)
Acronym: EROS+CP-Japan
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00093
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Retrospective; Real-World Effectiveness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- PROMPT: PATIENTS INITIATING BGF WITHIN 30-DAYS OF EXACERBATION
  Interventions: Drug: BGF
- DELAYED: PATIENTS INITIATING BGF WITHIN 31-180 DAYS OF EXACERBATION
  Interventions: Drug: BGF
- VERY DELAYED: PATIENTS INITIATING BGF BETWEEN 181 AND 365 DAYS AFTER EXACERBATION
  Interventions: Drug: BGF

INTERVENTIONS:
Drug: BGF — BUDESONIDE/GLYCOPYRRONIUM/FORMOTEROL

SUMMARY:
A retrospective real-world data study, assessing the relationship between the timing of Budesonide/Glycopyrrolate/Formoterol initiation following an exacerbation and the occurrence of subsequent exacerbations, severe cardiopulmonary events and other real-world outcomes in Japan

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (at any position) before or on the index date

  * 1 dispensation of BGF on or following the launch date of BGF in Japan
* Patients must have evidence of at least one qualifying COPD exacerbation event, which qualify the initiation of triple therapy. The exacerbation event must occur within the 12-month period preceding BGF initiation and on or after BGF launch in Japan (i.e., 04 September 2019). The earliest qualifying COPD exacerbation event will be set as the index date.

  * 12 months of continuous health plan enrollment preceding the qualifying COPD exacerbation date
  * 1 day of continuous enrollment following the qualifying COPD exacerbation date
* Age ≥ 40 years on the qualifying COPD exacerbation date

Exclusion Criteria:

* Presence of ≥ 2 records of respiratory cancer diagnoses occurring at least 1 month apart during the 12-month baseline period preceding the qualifying COPD exacerbation or during the follow-up period
* Presence of ≥ 1 dispensation of SITT during the 12-month baseline period preceding the index date through BGF initiation
* Patients who only have 1 moderate COPD exacerbation in 12-months period prior to BGF initiation with no dispensation of long-acting inhaled COPD maintenance treatment during the 12-months baseline period preceding the qualifying COPD exacerbation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The overall study population will include adult patients (aged ≥ 40) with COPD in Japan who have experienced a qualifying COPD exacerbation (defining the index date) on or after the BGF launch in Japan (i.e., 04 September 2019) for which triple therapy (i.e., BGF) could have been initiated per local or global guidelines
Sampling Method: Non-Probability Sample
Enrollment: 3402 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Annualized COPD Exacerbation Event Rate | Annualized rates from index exacerbation through end of data availability; median follow-up 713 days
  Annualized rates of COPD exacerbation events observed from index date (qualifying exacerbation event) through study completion (or until end of data availability with a median follow-up of 713 days

SECONDARY OUTCOMES:
Annualized Cardiopulmonary Event Rate | Annualized rates from index exacerbation through end of data availability with median follow-up of 713 days
  Annualized rates of cardiopulmonary events observed from index date (qualifying exacerbation event) through study completion (until end of data availability) with median follow-up time of 713 days.

OTHER OUTCOMES:
Time to and rate of all-cause mortality | Annualized incidence of mortality from index exacerbation through end of data availability; median follow-up 713 days
  Annualized incidence of all-cause mortality observed from index date (qualifying exacerbation event) through study completion (until end of data availability with median follow-up time of 713 days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pollack, MS, Study Director — AstraZeneca
Locations (1):
- AstraZeneca, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D5980R00093_CSR synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00093&attachmentIdentifier=08b65846-4caf-4f04-9f2f-081349e20a1b&fileName=D5980R00093_CSR_synopsis_Redacted.pdf&versionIdentifier=